CLINICAL TRIAL: NCT05945862
Title: Comprehensive Training Program to Promote Healthy Lifestyles and Prevent Food Insecurity and Child Malnutrition in Communities From the Yaqui Valley, Mexico
Brief Title: Healthy Lifestyle Promotion Program in Communities From the Yaqui Valley
Acronym: NUTRIGANDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Tecnologico de Sonora (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, ANA MARIA RENTERIA MEXIA, PhD, Instituto Tecnologico de Sonora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LNPAS_002
Record Dates: First submitted 2023-06-21; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2
Keywords: Healthy lifestyle intervention; Cardiovascular Disease Prevention; Mother-Child intervention
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Health Promotion and Disease Prevention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition-Physical activity Program (Experimental): Participants within the nutrition education and physical activity program
  Interventions: Behavioral: NUTRIGANDO

INTERVENTIONS:
Behavioral: NUTRIGANDO — Program consisting in nutrition education and physical activity training to promote healthy lifestyles

SUMMARY:
The aim is to evaluate the change in indicators of lifestyle and its effect on cardiometabolic biomarkers as a response to an integrative mother-child intervention to promote healthy lifestyles and prevent food insecurity and child malnutrition in vulnerable communities in the Yaqui Valley, Sonora, Mexico. The intervention consists in a program including nutrition education and physical activity training, with a total duration of 6 months. The proposal addresses the problem in an integrative and non-conventional way, generating new multifactorial knowledge of cardiometabolic and behavioral markers, and their relationship with each other, helping to reduce family food insecurity and improving lifestyle and health, and to support vulnerable families in achieving social justice in the field of nutrition.

DETAILED DESCRIPTION:
At present, the development and implementation of interventions in low-income families linking child malnutrition and food insecurity with cardiometabolic diseases, which are fundamental national health problems, is a priority. Educating mothers in this context is a fundamental tool for the prevention and early detection of nutritional diseases, since they are the main caregivers at home, and play a unique role as agents of change and promoters of family well-being. In addition, by training a child in healthy lifestyles, a healthy adult is being developed for the future, who in turn will raise healthy families. The aim of the study is to evaluate the change in indicators of lifestyle, such as diet and physical activity, and its effect on cardiometabolic biomarkers in response to an integrative mother-child intervention to promote healthy lifestyles and to prevent food insecurity and child malnutrition in vulnerable communities in the Yaqui Valley in Sonora, Mexico. The intervention consists in promoting healthy lifestyles for mothers and children in a 6-month program including: food-nutrition education to prevent child malnutrition and cardiometabolic diseases, promotion of planned physical activity, education for child health and cooking workshops. The proposal aims to address the problem in an integrative and non-conventional way, generating new knowledge from the multifactorial field of family, cardiometabolic and behavior, and it will be carried out in vulnerable rural communities. The culture and traditions of the region will be considered in the intervention so that families empower themselves and manage to develop and adopt healthy lifestyles within home, and thereby influencing the well-being and social justice of vulnerable communities. The proposal entails the participation of the mother-child dyad, evaluating the basal risk conditions, and the subsequent change in response to the intervention. This family intervention represents a sustainable community model that incorporates health and combats food insecurity.

ELIGIBILITY:
Inclusion Criteria:

* Children: ages 7 to 12 years.
* Parents: father, mother or guardian, all adults.
* Residency in Yaqui Valley, Sonora, Mexico.
* Show interest and time availability to complete all the protocol and measurements.

Exclusion Criteria:

* Children whose parents have not signed the informed consent.
* Those with cardiometabolic diseases such as diabetes, hypertension, etc. and therefore are subjected to a specific diet or therapeutic treatment.
* Those with any mental condition or illness, as well as any condition that includes a specific diet, exercise and/or lifestyle treatment/therapy that it would not reflect the common habits.
* Others: any other condition that physically affects the ability to participate in the program

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2023-08-11 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | 6 months
  Weight in kg measured by a portable body composition scale
Height | 6 months
  Height in cm measured by a portable stadiometer
Body fat | 6 months
  Body fat in kg measured by a portable body composition scale
Body mass index | 6 months
  Body mass index (BMI) calculated from weight divided by height (in squared meters)
Waist circumference | 6 months
  Waist circumference in cm using a Lufkin tape
Blood pressure | 6 months
  Systolic and diastolic blood pressure measured with a blood pressure monitor
Physical activity | 6 months
  Physical activity will be measured using the International Physical Activity Questionnaire, which measures the time per week spent on vigorous, moderate, light, and sedentary physical activities.
Fasting glucose | 6 months
  Measured in serum using a clinical chemistry analyzer
Total cholesterol | 6 months
  Measured in serum using a clinical chemistry analyzer
Triglycerides | 6 months
  Measured in serum using a clinical chemistry analyzer

SECONDARY OUTCOMES:
Psychosocial well-being | Baseline
  Psychosocial well-being in children measured using the Strengths and Difficulties Questionnaire (SDQ) for parents, which asks about positive and negative attributes across next characteristics: Total difficulties (scale from 0 to 40, highest is the worse); Emotional symptoms (scale from 0 to 10, highest is the worse); Conduct problems (scale from 0 to 10, highest is the worse); Hyperactivity/Inattention (scale from 0 to 10, highest is the worse); Peer Relationship Problems (scale from 0 to 10, highest is the worse); and Prosocial Behavior (scale from 0 to 10, lower is the worse).
Family interaction | Baseline
  Measured through The McMaster Family Assessment Device (FAD), which is a 60-item questionnaire that measures an individual's perceptions of his/her family. The score is calculated by adding the responses (1-4) for each scale and dividing by the number of items in each scale (6-12). Higher scores indicate worse levels of family functioning.
Traditional Mexican Diet Score | 6 months
  Foods within the Traditional Mexican Diet by the score proposed by Valerino-Perea et al. (2021), which consists of a score from a minimum of 0 to a maximum of 21, in which 21 is the best score for the Traditional Mexican Diet
Food intake | 6 months
  Food intake measured by duplicated 24 hour recalls
Lifestyle | 6 months
  Measured by the Fantastic questionnaire that includes the dimensions: F = Family and friends (2 items); A = Activity and Associativity (3 items); N = Nutrition (3 items); T = Tobacco (2 items); A = Alcohol and other substances (6 items); S = Sleep and stress (3 items); T = Type of personality (3 items); I = Introspection (3 items); and C = Control of health (3 items). The score ranges from 0 to 50, with the highest score being the best (a healthy lifestyle).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Renteria Mexia, PhD, Principal Investigator — Instituto Tecnologico de Sonora
Locations (1):
- Instituto Tecnologico de Sonora, Ciudad Obregón, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez-Cordero S, Cuevas-Nasu L, Moran-Ruan MC, Mendez-Gomez Humaran I, Avila-Arcos MA, Rivera-Dommarco JA. Overweight and obesity in Mexican children and adolescents during the last 25 years. Nutr Diabetes. 2017 Mar 13;7(3):e247. doi: 10.1038/nutd.2016.52. PMID 28287630
- [Background] Barquera S, White M. Treating Obesity Seriously in Mexico: Realizing, Much Too Late, Action Must Be Immediate. Obesity (Silver Spring). 2018 Oct;26(10):1530-1531. doi: 10.1002/oby.22296. No abstract available. PMID 30277025
- [Background] Tonnies T, Rathmann W, Hoyer A, Brinks R, Kuss O. Quantifying the underestimation of projected global diabetes prevalence by the International Diabetes Federation (IDF) Diabetes Atlas. BMJ Open Diabetes Res Care. 2021 Aug;9(1):e002122. doi: 10.1136/bmjdrc-2021-002122. No abstract available. PMID 34400463
- [Background] Swinburn BA, Kraak VI, Allender S, Atkins VJ, Baker PI, Bogard JR, Brinsden H, Calvillo A, De Schutter O, Devarajan R, Ezzati M, Friel S, Goenka S, Hammond RA, Hastings G, Hawkes C, Herrero M, Hovmand PS, Howden M, Jaacks LM, Kapetanaki AB, Kasman M, Kuhnlein HV, Kumanyika SK, Larijani B, Lobstein T, Long MW, Matsudo VKR, Mills SDH, Morgan G, Morshed A, Nece PM, Pan A, Patterson DW, Sacks G, Shekar M, Simmons GL, Smit W, Tootee A, Vandevijvere S, Waterlander WE, Wolfenden L, Dietz WH. The Global Syndemic of Obesity, Undernutrition, and Climate Change: The Lancet Commission report. Lancet. 2019 Feb 23;393(10173):791-846. doi: 10.1016/S0140-6736(18)32822-8. Epub 2019 Jan 27. No abstract available. PMID 30700377
- [Background] Valerino-Perea S, Armstrong MEG, Papadaki A. Development of an index to assess adherence to the traditional Mexican diet using a modified Delphi method. Public Health Nutr. 2021 Oct;24(14):4387-4396. doi: 10.1017/S1368980020004565. Epub 2020 Nov 13. PMID 33183382